CLINICAL TRIAL: NCT03377595
Title: Post-cesarean Section Analgesic Safety and Efficacy of EXPAREL (Liposomal Bupivacaine) Infiltration Locally Versus Transversus Abdominis Plane Infiltration
Brief Title: Post C-Section Pain Control Using EXPAREL
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of resources, no data collected
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OBGYN-2017-26339
Record Dates: First submitted 2017-12-01; First posted 2017-12-19 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TAP (Transversus Abdominis Plane) block (Experimental): 20-mL dose of EXPAREL 266 mg expanded in volume with 20 mL normal saline plus 20 mL 0.25% bupivacaine for a total volume of 60 mL m.A 2-point classic TAP block will be performed under ultrasound guidance within 1 hour (± 30 minutes) following skin incision closure of the C-section.
  Interventions: Drug: Exparel
- Wound infiltration (Experimental): 20 mL of EXPAREL 266 mg expanded in volume with 40 mL normal saline for a total volume of 60 mL, infiltrated in the fascia prior to skin closure with attention to infiltrate the angles of the incision.
  Interventions: Drug: Exparel

INTERVENTIONS:
Drug: Exparel — TAP (Transversus Abdominis Plane) block
  Other Names: Saline
  Arms: TAP (Transversus Abdominis Plane) block
Drug: Exparel — Wound infiltration
  Other Names: Saline
  Arms: Wound infiltration

SUMMARY:
Evaluating the safety and efficacy of EXPAREL (Liposomal Bupivacaine ) for pain control in patients undergoing scheduled cesarean section by giving it either as infiltration in Transversus Abdominis Plane after finishing the procedure or through wound infiltration into the fascia prior to closure of skin

ELIGIBILITY:
Inclusion Criteria:

1. Females 18 years of age and older at screening.
2. Term pregnancies of 37 to 42 weeks gestation, scheduled to undergo elective C-section.
3. ASA (American Society of Anesthesiologists) physical status 1, 2, or 3 are able to provide informed consent, adhere to the study visit schedule, and complete all study assessments

Exclusion Criteria:

1. Age <18
2. BMI > or equal to 40 or otherwise not anatomically appropriate to undergo a TAP block.
3. Planned general anesthetic
4. Cesarean delivery via vertical skin incision
5. Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications.
6. Planned concurrent surgical procedure with the exception of salpingo-oophorectomy or tubal ligation.
7. Severely impaired renal or hepatic function (eg, serum creatinine level >2 mg/dL [176.8 µmol/L], blood urea nitrogen level >50 mg/dL [17.9 mmol/L], serum aspartate aminotransferase [AST] level >3 times the upper limit of normal , or serum alanine aminotransferase [ALT] level >3 times the upper limit of normal.)
8. Subjects at an increased risk for bleeding or a coagulation disorder (defined as platelet count less than 80, 000 × 103/mm3 or international normalized ratio greater than 1.5).
9. Concurrent painful physical condition that may require analgesic treatment (such as long-term, consistent use of opioids) in the postsurgical period for pain that is not strictly related to the surgery and which may confound the postsurgical assessments.
10. Clinically significant medical disease in either the mother or baby that, in the opinion of the investigator, would make participation in a clinical study inappropriate. This includes any psychiatric or other disease in the mother that would constitute a contraindication to participation in the study or cause the mother to be unable to comply with the study requirements.
11. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
12. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study
13. Previous participation in an EXPAREL study.
14. Any clinically significant event or condition uncovered during the surgery (eg, excessive bleeding, acute sepsis) that might render the subject medically unstable or complicate the subject's postsurgical course.
15. Initiation of treatment with any of the following medications within 1 month of study drug administration or if the medication(s) are being given to control pain: selective serotonin reuptake inhibitors (SSRIs), selective norepinephrine reuptake inhibitors (SNRIs), gabapentin, pregabalin (Lyrica®), or duloxetine (Cymbalta®). If a subject is taking one of these medications for a reason other than pain control, she must be on a stable dose for at least 1 month prior to study drug administration.
16. Use of any of the following medications within the times specified before surgery: long-acting opioid medication, non-steroidal anti-inflammatory drugs (NSAIDs), or aspirin (except for low-dose aspirin used for cardioprotection) within 3 days, or any opioid medication or acetaminophen within 24 hours.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption | 72 hours
  Total opioid medication use by patient after having cesarean section

SECONDARY OUTCOMES:
Time to first rescue opioid pain medication | 72 hours
  Time till the patient asks for opioid medication for breakthrough pain
Percentage of opioid-free subjects | 24,48, and 72 hours
  Percentage of patients didn't require any opioid medications after the cesarean section
Patient's satisfaction | through 72 hours post-op or at discharge
  Patient's satisfaction questionnaire with pain control
VAS (visual analogue scale) pain scores | at 6, 12, 18, 24, 30, 36, 42, 48, and 72 hours after surgery
  pain level assessment using visual assessment pain score which ranges from zero for no pain to 10 intolerable pain
Number of participants with EXPAREL related adverse events | through day 14 post-op
  side effects of EXPAREL
Allergic reactions attributable to local anesthetic use | through day14 post-op
  Such as allergies, rash etc...
Wound complications | through day 14 post-op
  cesarean section wound complications like infection, hematoma, and dehiscence

CONTACTS AND LOCATIONS:
Overall Officials: Hiba Mustafa, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No